CLINICAL TRIAL: NCT02490657
Title: Effects of Iloprost on Pulmonary Hemodynamics and Oxygenation in Patients of Chronic Obstructive Pulmonary Disease During One-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 4-2015-0283
Record Dates: First submitted 2015-06-15; First posted 2015-07-07 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Video-assisted Thoracoscopic Surgery; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iloprost group (Experimental)
  Interventions: Drug: Inhaled iloprost
- normal saline (Placebo Comparator)
  Interventions: Drug: normal saline (Saline 0.9%)

INTERVENTIONS:
Drug: Inhaled iloprost — Nebulized agents (Iloprost or normal saline) were randomized by computer-generated randomization. The patients and anesthesiologist, who administered inhalation and conducted all this trial, were blinded to the medication allocation. An anesthesiologist, who responsible for preparation of medication, was the only person recognizing of the randomization code during trial.
  Enrolled patients were received 20 μg iloprost or placebo (norma saline). Iloprost was diluted in normal saline to obtain 2ml solution. Control group were inhaled comparable dose of normal saline. Iloprost or normal saline was inhaled through an ultrasonic nebulized system in inspiratory limb.
  Arms: Iloprost group
Drug: normal saline (Saline 0.9%)
  Arms: normal saline

SUMMARY:
The inhaled Iloprost, approved for pulmonary hypertension, caused increase in oxygenation, and increase exercise tolerance in ARDS or chronic obstructive pulmonary disease. Inhaled iloprost has been researched in animal study, but not yet in human during one-lung ventilation. The investigators will enroll patients who diagnosed moderate to severe chronic obstructive pulmonary disease, preoperative pulse oximetry (SpO2) of below 95% at room air or PaO2 /FiO2 ratio< 150 mmHg after initiating one-lung ventilation. The primary outcome is pulmonary oxygenation expressed by PaO2 /FiO2 ratio. And secondary outcome is assessment of cardiac function including Tei-index during nebulizing iloprost. The investigators hypothesized inhaled iloprost will improve oxygenation and decrease the FiO2 in chronic obstructive pulmonary disease during one-lung ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic obstructive pulmonary disease was defined as FEV1/FVC ratio < 0.7 and an FEV 1 of 80% or less after inhalation bronchodilator : 1. Above 40 years of age.
2. American Society of Anesthesiologists (ASA) Physical Status II, III.
3. Preoperative SpO2 95 % or less at room air (spontaneous ventilation) or 4. PaO2 /FiO2 ratio< 150 mmHg after initiating one-lung ventilation

Exclusion Criteria:

1. Severe functional liver or kidney disease
2. Diagnosed HF (LV ejection fraction <50% , or wall motion abnormality)
3. Arrhythmia or received treatment with antiarrythmic drug .
4. Severe bradycardia(HR < 45 bpm) and AV block 6. pathologic esophageal lesion (esophageal stricture or varix ) 7. pregnancy 8. PaO2 /FiO2 ratio ≥ 150 mmHg after initiating one-lung ventilation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
PaO2 /FiO2 ratio during one-lung ventilation | oxygenation changes from baseline (OLV), in 30 min after nebulizing iloprost or normal saline(ILO-30), in 60 min after nebulizing iloprost or normal saline(ILO-60), to after 20 min in postanaestheticcare unit(PACU)

SECONDARY OUTCOMES:
biventricular diastolic function | biventricular diastolic function changes from baseline(baseline), 60 min after nebulizing iloprost or normal saline (ILO)
  E/e' estimated by tissue Doppler index

OTHER OUTCOMES:
Tei-index (tissue Doppler image-derived myocardial performance ) at lateral and septal | myocardial performance changes from baseline(baseline), 60 min after nebulizing iloprost or normal saline (ILO)
  Tei-index (tissue Doppler image-derived myocardial performance ) at lateral and septal

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, Seoul, South Korea